CLINICAL TRIAL: NCT03363308
Title: Effects of a Health Workforce Capacity Building and Quality Improvement Intervention on Intrapartum Stillbirth, Early Newborn Mortality and Post-pregnancy Family Planning in Kinshasa: a Cluster Randomized Evaluation
Brief Title: Effects of a Health Workforce Capacity Building and Quality Improvement Intervention in Kinshasa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1156220
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Maternal Death; Infant Death; Stillbirth
MeSH Terms: conditions — Maternal Death; Infant Death; Stillbirth | interventions — Data Collection; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized trial in phase I and interrupted time series in phase II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): training for health care workers supplemented by QI teams
  Interventions: Behavioral: training for health care workers supplmented by QI teams
- Phase 2 (No Intervention)

INTERVENTIONS:
Behavioral: training for health care workers supplmented by QI teams — Jhpiego will deliver maternal and newborn health and family planning (MNH+FP) training using evidence-based low-dose, high-frequency (LDHF) learning approaches and support hospital staff-led quality improvement efforts to increase the coverage of facility-based high-impact interventions, including care of the mother and newborn on the day of birth and through the first week postpartum and post abortion services.
  Other Names: Practice coordinator training after training session; Practice sessions using anatomic models; SMS reminder messages and quizzes; Routine calls between mentors and providers; Health information officer training; Data collection and use training; Supply of simulators, equipment, kits and other; Develop quality improvement teams and review of action plans; Routine calls between project staff and mentors
  Arms: Phase 1

SUMMARY:
The aim of the study is to evaluate a health workforce capacity building and quality improvement intervention focused on integrated day-of-birth and post-pregnancy care at 16 hospitals in Kinshasa, Democratic Republic of Congo. The intervention package consists of a low-dose, high-frequency (LDHF) training of health workers, support for quality improvement teams, and provision of critical equipment, supplies and drugs within a quality improvement (QI) framework.

DETAILED DESCRIPTION:
The health workforce capacity building and quality improvement intervention will be implemented in two phases: eight facilities will receive the intervention in phase 1 and the remaining eight facilities will receive the intervention in phase 2.

Objective 1: For objective 2 on facility-based health outcomes, the study design is a cluster-randomized evaluation in phase 1. The intervention's effects will be assessed by comparing an intervention group and a control group of facilities. These will be selected from 16 Kinshasa health facilities. Intervention and control facilities' monthly reported health outcomes will be compared in a 12-month baseline period and 12-month period during and after the intervention implementation (Phase 1) in a difference-in-difference analysis. In Phase 2, all facilities will have their monthly service statistics and health outcomes reviewed for trends in improvement.

Overall, in Phase 1, eight intervention sites will be matched to eight sites serving as controls. In Phase 2, the eight Phase 1 control sites will then receive the same package as the intervention sites in Phase 1. Sites will be stratified by case load, low and high (over 90 births per month), and funding (public or private funding). Within each stratum, prior to start of the intervention, there will be random selection to intervention and control groups to allow for baseline comparability between groups.

ELIGIBILITY:
Inclusion Criteria:

* Health providers:

  * Currently on the roster of maternity ward providers working at one of the 16 selected facilities at the time of the training module.
  * Willing to attend a Jhpiego clinical training workshop and offer consent as study participant.
  * Age 18 or older.

Exclusion Criteria:

* there are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mean number or percent of items correctly answered | 1 day
  Each observed structured clinical exam (OSCE) or knowledge tests has between 13 and 38 items. A participant needs to achieve 85% correct score to pass at post-training to assess provider competencies. The main indicator for analysis will be the mean number of items (or percent of items) correctly answered. This mean percent of items correctly answered will be done pre-training, post-training and after 6 months. This will be done in the 8 intervention group facilities only in Phase I and again in the 8 new facilities in Phase II.
Intrapartum perinatal death ratio | 1 day
  Defined as death of a fetus during labor who had heart tones documented on arrival in the maternity and neonatal deaths prior to 24 hours, divided by total births.
Percent of women after childbirth who adopt a family planning method immediately post-pregnancy or intend to adopt a method by six weeks post-pregnancy. | 3 days
  Percent of women after childbirth who adopt a family planning method over all women who give birth in a facility

SECONDARY OUTCOMES:
maternal mortality | 3 days
  number of maternal deaths over number of live births

CONTACTS AND LOCATIONS:
Overall Officials: Virgile Kikaya, Principal Investigator — Jhpiego DRC
Locations (1):
- Jhpiego DRC, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No